CLINICAL TRIAL: NCT01398384
Title: The Effects of Nitric Oxide for Inhalation on Myocardial Infarction Size
Brief Title: Effects of Nitric Oxide for Inhalation in Myocardial Infarction Size
Acronym: NOMI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LCC2010.01
Record Dates: First submitted 2011-07-18; First posted 2011-07-20 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Acute Myocardial Infarction
Keywords: ST Elevation MI; STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Nitric Oxide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nitric Oxide (Active Comparator): nitric oxide for inhalation
  Interventions: Drug: Nitric Oxide
- Placebo (Placebo Comparator): inhalation gas
  Interventions: Drug: MI size at 48-72 hours

INTERVENTIONS:
Drug: Nitric Oxide — MI size at 48-72 hours
  Other Names: vasoKINOX 450
  Arms: Nitric Oxide
Drug: MI size at 48-72 hours — Placebo gas
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effects of Nitric Oxide for Inhalation on Myocardial Infarction Size.

DETAILED DESCRIPTION:
The primary objective of the trial is to assess whether or not inhaled nitric oxide can decrease myocardial infarction (MI) size as a fraction of left ventricular size at 48-72 hours in patients presenting with an ST segment elevation MI who undergo successful percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Acute myocardial infarction (defined as an episode of chest pain or related symptom lasting greater than 2 hours but less than 12 hours and electrocardiographic evidence of ST elevation (measured as 0.08 seconds after the J point; sum greater or equal to 0.6 mV in leads I, II, III, AVL, AVF, V1-V6).
2. No evidence of congestive heart failure (no S3 or evidence of pulmonary edema) and normal oxygen saturation on ≤ 2L oxygen by NC.
3. All patients must undergo successful percutaneous coronary intervention for TIMI 0 or 1 coronary flow with resulting TIMI 2 or 3 (residual stenosis less than 30% if stented and less than 50% if opened by balloon angioplasty).
4. Age > 18 years.
5. Signed EC approved informed consent.

Exclusion Criteria:

1. Prior myocardial infarction (as determined by patient history and/or ECG), cardiac surgery, or severe pericardial, congenital, cardiomyopathic or valvular heart disease.
2. Requirement for urgent cardiac surgery.
3. Previous CABG or PCI.
4. Left bundle branch block.
5. Unable to tolerate magnetic resonance imaging (including disallowed metallic implants or BMI > 35) or unable to tolerate gadolinium contrast media, including patients with calculated creatinine clearance less than 60 ml/min/1.73 m2 BSA.
6. Active or recent hemorrhage requiring an invasive procedure for evaluation or transfusion within 6 weeks prior to presentation or hemorrhagic stroke within the 6 weeks prior to presentation.
7. Known or suspected aortic dissection.
8. Prior history of pulmonary disease requiring chronic oxygen therapy.
9. Pregnancy, lactating and woman of childbearing potential.
10. Use of investigational drugs or device within the 30 days prior to enrollment to the study. Investigational uses of approved therapies will be allowed.
11. Medical problem likely to preclude completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2010-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Myocardial infarction size as a fraction of left ventricular size | 48-72 hours
  Myocardial infarction size as a fraction of left ventricular size at 48-72 hours in patients presenting with an ST segment elevation MI who undergo successful percutaneous coronary intervention.

SECONDARY OUTCOMES:
MI size, extent and transmurality of microvascular obstruction | 48-72 hours
  MI size, extent and transmurality of microvascular obstruction measured by MRI
MI size normalized to area at risk | 48-72 hours
Myocardial perfusion at coronary angiography at the completion of PCI (corrected TIMI frame count and myocardial blush grade). | at completion of PCI, as expected 1 day
Transmurality of infarct (as average percent wall thickness in all segments showing delayed enhancement). | at 48 - 72 hours and 4 months
Myocardial perfusion(MRI). | at 48-72 hours and 4 months
Global and regional left ventricular function and left ventricular mass at 48 - 72hours and 4 months after MI and the change in global LV function and mass between 48-72 hours and 4 months. MI size as a fraction of LV size at 4 months after MI. | 48-72 hours and 4 months
Resolution of ST segment elevation (serial ECGs) as indicated by the decrease in the total ST elevation (in mV) at 4 hours compared with that observed at enrollment. | at 4 hours
Troponin T levels and CPK-MB area under the curve at 48 hours. | 48 hours
Change in adverse remodeling parameters (compared with 48-72 hours):changes in LV end-diastolic volume, end-systolic volume, end-diastolic myocardial wall thickness in infarct, peri-infarct and remote areas and in sphericity index. | 4 months
  Change in adverse remodeling parameters (compared with 48-72 hours):changes in LV end-diastolic volume, end-systolic volume, end-diastolic myocardial wall thickness in infarct, peri-infarct and remote areas and in sphericity index at end-diastole and end-systole.
Death, nonfatal recurrent MI, recurrent ischemia necessitating re-hospitalization, PCI, or surgical revascularization, and stroke (i.e. combined CV endpoint) at 4 months. Enzyme leak during subsequent scheduled PCI will not be considered new ischemia/MI. | 4 months
Assess the safety of inhaled NO for this use as determined by reported adverse events (including bleeding and laboratory changes). | during treatment gas period, an average of 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Janssens, Prof Dr, Principal Investigator — UZ Leuven; Frans Van de Werf, Prof Dr, Principal Investigator — UZ Leuven
Locations (4):
- Belgium (2):
  - Jessa Hospital, Hasselt
  - UZ Leuven, Leuven
- Semmelweis University Heart Center, Budapest, Hungary
- John Paul II Hospital, Krakow, Poland

REFERENCES:
- [Derived] Janssens SP, Bogaert J, Zalewski J, Toth A, Adriaenssens T, Belmans A, Bennett J, Claus P, Desmet W, Dubois C, Goetschalckx K, Sinnaeve P, Vandenberghe K, Vermeersch P, Lux A, Szelid Z, Durak M, Lech P, Zmudka K, Pokreisz P, Vranckx P, Merkely B, Bloch KD, Van de Werf F; NOMI investigators. Nitric oxide for inhalation in ST-elevation myocardial infarction (NOMI): a multicentre, double-blind, randomized controlled trial. Eur Heart J. 2018 Aug 1;39(29):2717-2725. doi: 10.1093/eurheartj/ehy232. PMID 29800130